CLINICAL TRIAL: NCT05260099
Title: Post Market Clinical Follow up (PMCF) Medical Device (MD) Registry of the Alteco® LPS Adsorber to Remove Lipopolysaccharide (LPS) in Patients With Suspected Endotoxemia, With Severe Symptom(s)/Complication(s) and Their Stabilization Outcomes: REMOVE LPS Registry
Brief Title: Remove LPS Registry
Status: Withdrawn | Type: Observational
Why Stopped: Company decision not to start study
Sponsor: Alteco Medical AB (Industry)
Responsible Party: Sponsor
Other Study IDs: Remove LPS Registry
Record Dates: First submitted 2022-02-18; First posted 2022-03-02 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Suspected or Diagnosed Endotoxemia Casued by Gram-negative Bacteria

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective: Patients not treated with LPS Adsorber
- Prospective: Patients treated with LPS Adsorber
  Interventions: Device: LPS Adsorber

INTERVENTIONS:
Device: LPS Adsorber — LPS Adsorber, binding endotoxin caused by suspected or verified gram-negative bacteria.
  Groups: Prospective

SUMMARY:
This registry will collect and validate regulatory-grade real-world data (RWD) on the usage of the LPS-Adsorber and the outcomes from using the LPS-Adsorber in various patient populations (various sub-registries) that also have suspected endotoxemia. This data can be then used in real-world evidence (RWE) generation. It will also create reusable infrastructure to allow creation or affiliation with many additional RWD/RWE efforts both prospective and retrospective in nature.

ELIGIBILITY:
Inclusion Criteria:

* Weight > 30 kilos

Specific sub-registry criteria are possible.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected or diagnosed sepsis caused by gram-negative bacteria.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-11 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint will be the time needed to achieve patient stabilization from the time of treatment. | 30 days

SECONDARY OUTCOMES:
Secondary Outcomes will be to document the change in a patient's symptoms of infection over time. | 30 days
Rate of complaints and incidents related to the medical device during the whole registry. | 30 days

IPD SHARING:
Plan to Share IPD: No